CLINICAL TRIAL: NCT05143229
Title: Phase I Trial Of Alpelisib Plus Sacituzumab Govitecan In Patients With Metastatic Or Locally Recurrent HER2-Negative Breast Cancer
Brief Title: Alpelisib And Sacituzumab Govitecan For Treatment Of Breast Cancer
Acronym: ASSET
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Priyanka Sharma, Principal Investigator, University of Kansas Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2021-ASSET
Record Dates: First submitted 2021-11-19; First posted 2021-12-03 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: HER2-negative; Metastatic/locally advanced; Sacituzumab govitecan; Alpelisib; RP2D; Trop-2 antibody-drug conjugate; PI3K inhibitor
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Alpelisib; sacituzumab govitecan

STUDY DESIGN:
Intervention Model Description: Standard 3+3 dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose level 1: alpelisib 250 mg plus sacituzumab govitecan 8 mg/kg (Experimental): Alpelisib: 250 mg by mouth daily Sacituzumab govitecan: 8 mg/kg intravenous on days 1 and 8 of each 21 (+/-2) day cycle
  Interventions: Drug: Alpelisib; Drug: Sacituzumab govitecan
- Dose level 2: alpelisib 250 mg plus sacituzumab govitecan 10 mg/kg (Experimental): Alpelisib: 250 mg by mouth daily Sacituzumab govitecan: 10 mg/kg intravenous on days 1 and 8 of each 21 (+/-2) day cycle
  Interventions: Drug: Alpelisib; Drug: Sacituzumab govitecan
- Dose level 3: alpelisib 300 mg plus sacituzumab govitecan 10 mg/kg (Experimental): Alpelisib: 300 mg by mouth daily Sacituzumab govitecan: 10 mg/kg intravenous on days 1 and 8 of each 21 (+/-2) day cycle
  Interventions: Drug: Alpelisib; Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Alpelisib — PI3K inhibitor
  Other Names: Piqray
Drug: Sacituzumab govitecan — Trop-2-directed antibody and topoisomerase inhibitor drug conjugate
  Other Names: Trodelvy

SUMMARY:
This study evaluates the safety and efficacy of sacituzumab govitecan plus alpelisib for treatment of metastatic or locally recurrent HER2-negative breast cancer.

ELIGIBILITY:
Inclusion criteria:

1. Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
2. Males and females age ≥ 18 years
3. ECOG Performance Status 0 - 2 (See Appendix A)
4. Histologically proven HER2-negative breast cancer (per current ASCO-CAP guidelines); HER2-negative breast cancer includes hormone receptor-positive (estrogen receptor and/or progesterone receptor-positive) breast cancer and TNBC.
5. HER2-negative breast cancer that at the time of study entry is either stage III (locally advanced) disease not amenable to curative therapy, or stage IV disease. Histological confirmation of recurrent/metastatic disease is encouraged but not required if clinical evidence of stage IV disease is available.
6. Have measurable or evaluable disease.
7. Ability to swallow and retain oral medicines.
8. No limitations to number of prior chemotherapies or endocrine therapies for metastatic disease.
9. All patients should have received at least one line of chemotherapy and at least one line of hormonal therapy (where appropriate) in either the advanced or neo/adjuvant setting. Patients who are candidates for anti-PD-1 and/or anti-PD-L1 therapy should have received at least one line of anti-PD-1 and/or anti-PD-L1 therapy in either the advanced or neo/adjuvant setting.
10. Prior palliative radiation therapy to bony metastases is allowed. A minimum of 14 days between the end of radiation treatment and start of study treatment is required.
11. Participants with previously treated brain metastases must be free of central nervous system symptoms and be >21 days from treatment of brain metastases. CNS brain metastasis should be clinically stable at the time of screening, and participant is not receiving steroids and/or enzyme inducing anti-epileptic medications for brain metastases.
12. Participants must be >2 weeks or 5 half-lives (whichever is longer) from prior systemic chemotherapy for breast cancer AND should have recovered to Grade 1 or better (except alopecia and neuropathy) from related side effects of any prior antineoplastic therapy prior to study entry.
13. Women of childbearing potential must have a negative serum pregnancy test 24 hours prior to initiating treatment.
14. Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence or to use approved forms of contraception for the duration of study participation and for 6 months following completion of therapy.
15. Fasting plasma glucose ≤140 mg/dL or ≤7.8 mmol/L
16. HbA1c ≤6.4%
17. Absolute neutrophil count ≥ 1500/uL NOTE: Patients with established diagnosis of benign neutropenia are eligible to participate with ANC between 1000-1500 if in the opinion of treating physician the trial treatment does not pose excessive risk of infection to the patient.
18. Platelets ≥ 100,000/uL (no transfusion allowed within 2 weeks)
19. Hemoglobin > 9 g/dL (which may be reached by transfusion)
20. Total bilirubin within normal range or ≤ 1.5x institutional upper limit of normal (IULN) if liver metastases are present, or total bilirubin ≤ 3.0x IULN with direct bilirubin within normal range in patients with well-documented Gilbert's Syndrome, which is defined as presence of unconjugated hyperbilirubinemia with normal results from CBC (including normal reticulocyte count and blood smear), normal liver function test results and absence of other contributing disease processes at the time of diagnosis.
21. AST(SGOT)/ALT(SPGT) ≤ 2.5x IULN or ≤ 5x IULN if liver metastases are present
22. Serum creatinine ≤ 1.5x IULN
23. Creatinine clearance ≥ 35 mL/min using Cockcroft-Gault formula
24. Potassium within institutional normal limits
25. Magnesium within institutional normal limits
26. Calcium (corrected for serum albumin) within institutional normal limits or ≤grade 1 according to NCI-CTCAE version 4.03 if judged clinically not significant by the investigator
27. Serum amylase ≤ 2x IULN
28. Serum lipase within institutional normal limits
29. Albumin ≥ 2.5 g/dL

Exclusion criteria:

1. Simultaneously enrolled in any therapeutic clinical trial
2. Current or anticipating use of other anti-neoplastic or investigational agents while participating in this study
3. Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
4. Is pregnant or breastfeeding
5. Has a known allergic reaction to any excipient contained in the study drug formulation Active Grade 3 (per the NCI CTCAE, Version 5.0) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment.
6. Patient has previously been treated with sacituzumab govitecan or alpelisib.
7. Patient has a concurrent malignancy or malignancy within 3 years of study enrollment (with the exception of adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer, or curatively resected cervical cancer).
8. Diabetes mellitus type I, or uncontrolled type II based on fasting plasma glucose and HbA1c meeting either of the following:

   * Fasting plasma glucose >140 mg/dL or >7.8 mmol/L
   * HbA1c ≥6.5% Note: For patients with fasting plasma glucose ≥ 100 mg/dL and/or HbA1c ≥5.7% (i.e. threshold for pre-diabetes) at baseline, lifestyle changes according to American Diabetes Association guidelines were recommended
9. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
10. Patient is classified into Child-Pugh class B or C.
11. Patient has a known history of HIV infection (testing not mandatory).
12. Patient has active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV). In patients with a history of HBV or HCV, patients with a detectable viral load will be excluded.
13. Patient has symptomatic/untreated CNS disease.
14. Patient has active cardiac disease or a history of cardiac dysfunction including any of the following:

    * Uncontrolled hypertension defined by a systolic blood pressure (SBP) ≥ 160 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mm Hg, with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening.
    * Unstable angina pectoris within 6 months prior to study entry
    * Symptomatic pericarditis
    * Documented myocardial infarction within 6 months prior to study entry
    * Coronary artery bypass graft within 6 months prior to study entry
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
    * Documented cardiomyopathy
    * Patient has a left ventricular ejection fraction (LVEF) < 50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
    * Patient has any of the following cardiac conduction abnormalities:

      * Ventricular arrhythmias, except for benign premature ventricular contractions
      * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medicine
      * Conduction abnormality requiring a pacemaker
      * Other cardiac arrhythmia not controlled with medication
15. Patient has a QTcF > 470 msec if female and >450 msec if male on the screening ECG (using the QTcF formula).
16. Patient is currently receiving treatment with a medication that has a known risk to prolong the QT interval or induce Torsades de Pointes and the treatment cannot be discontinued or switched to a different medication prior to start of study drug.
17. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects.
18. Participant has received palliative radiation therapy ≤ 2 weeks prior to starting study drug, or has not recovered to grade 1 or better from related side effects of such therapy (with the exception of alopecia).
19. Patient is currently receiving or has received high-dose systemic corticosteroids (≥20mg of prednisone or its equivalent) ≤ 2 weeks prior to starting study drug or has not fully recovered from side effects of such treatment.

    Note: The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
20. Patient is currently receiving treatment with drugs known to be moderate or strong inhibitors or inducers of isoenzyme CYP3A. The patient must have discontinued strong inducers for at least one week before the start of treatment.
21. Patient is currently receiving treatment with inhibitor(s) of BCRP (see Appendix B, table with heading Prohibited BRCP inhibitors). The patient must have discontinued BCRP inhibitors for at least one week before the start of treatment.
22. Patient is currently receiving warfarin or other coumarin-derived anti-coagulant for treatment, prophylaxis or otherwise.
23. Patient has received previous treatment with a PI3K inhibitor or AKT inhibitor
24. Patient has a history of acute (within one year of study entry) pancreatitis or past medical history of chronic pancreatitis.
25. Patient has pneumonitis or interstitial lung disease.
26. Patient has unresolved osteonecrosis of the jaw.
27. Patient has inflammatory breast cancer.
28. Patient has a history of severe cutaneous reactions, such as Steven-Johnson Syndrome (SJS), erythema multiforme (EM), toxic epidermal necrolysis (TEM), or drug reaction with eosinophilia and systemic syndrome (DRESS).
29. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation in the clinical study (including, but not limited to: severe immune disease, certain degenerative diseases, certain other acute or chronic concurrent illnesses).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of alpelisib + sacituzumab govitecan | 21 days
  Standard 3+3 dose escalation design (three dose levels of alpelisib plus sacituzumab govitecan) with dose-limiting toxicities (DLT) assessed during the first treatment cycle. If two or more of the six patients experienced a dose-limiting toxicity, dosing escalation would cease and maximum tolerated dose (MTD) would be reached. RP2D was the next lower dose at which <1/6 subjects experienced a DLT.

SECONDARY OUTCOMES:
Pharmacokinetics of alpelisib when administered with sacituzumab govitecan | In cycle 1, from prior to sacituzumab govitecan dosing through 48 hours after sacituzumab govitecan dosing
  Alpelisib area under the curve (AUC): blood sampling pre-dose and 0.5, 1, 2, 3, 4, 6, 24, and 48 hours post-sacituzumab govitecan dose
Pharmacokinetics of sacituzumab govitecan when administered with alpelisib | In cycle 1, from prior to sacituzumab govitecan dosing through 48 hours after sacituzumab govitecan dosing
  Sacituzumab govitecan, free SN-38, and total SN-38 area under the curve (AUC): blood sampling pre-dose and 0.5, 1, 2, 3, 4, 6, 24, and 48 hours post-sacituzumab govitecan dose
Overall response rate (ORR) in patients with measurable disease | From start of study treatment until removal from study treatment; estimated 24 months maximum.
  ORR includes complete response (CR) plus partial response (PR). As evaluated per RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Sharma, MD, Principal Investigator — University of Kansas Medical Center
Locations (7):
- United States (7):
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - The University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - The University of Kansas Cancer Center - Indian Creek, Overland Park, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - The University of Kansas Cancer Center - North Kansas City Hospital, Kansas City, Missouri
  - The University of Kansas Cancer Center - North, Kansas City, Missouri
  - The University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri